CLINICAL TRIAL: NCT07100522
Title: Clinical Evaluation of the Nuance Audio Hearing Aid in Adults With Mild to Moderate Hearing Difficulties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luxottica Group S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C24.08
Record Dates: First submitted 2025-05-15; First posted 2025-08-03 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Hearing Impairment
Keywords: Nuance Audio hearing device, speech in noise, hearing difficulties; mild to moderate
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Intervention Model Description: post-market interventional, usability
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Clinical performance speech intelligibility with Hearing aid in spectacle frame form factor (Other): This study uses a within-subjects design in which participants complete assessments in both unaided and aided conditions, using the Nuance Audio Glasses as the investigational hearing aid device. Each participant attends two sessions at the National Acoustic Laboratories (NAL), with testing conducted in controlled and real-world environments.
  Research methods include:
  Audiometric assessments: Pure-tone audiometry, tympanometry, and Real Ear Measurements (REMs).
  Speech perception testing: Conducted in both quiet and noise using validated Australian English BKB sentence materials.
  Real-world assessments: Moderated walking tour in various acoustic settings (e.g., quiet rooms, traffic noise, multi-talker babble).
  Self-reported measures: Questionnaires assessing hearing difficulty (HHIE-S), listening goals (COSI), perceived benefit (IOI-HA), and device preference and satisfaction.
  Interventions: Device: Hearing aid in spectacle frame form factor; Device: hearing aid

INTERVENTIONS:
Device: Hearing aid in spectacle frame form factor — eyewear frames embedded with groundbreaking technology which seamlessly integrate an air conduction hearing aid (over-the-counter "OTC", in the United States) intended to amplify sound for adult users (18yrs and older) with a perceived mild to moderate hearing impairment. Nuance Audio Glasses may, if necessary, be used in association with prescription lenses for those adults who also require correction of visual defects. Nuance Audio Glasses can be worn all day and can be easily configured via the App to adapt to any situation, from business meetings to family time.
Device: hearing aid — Hearing aid in spectacle frame form factor

SUMMARY:
The research will produce clinical effectiveness performance metrics using standardised procedures of the Nuance Audio hearing device.

DETAILED DESCRIPTION:
EssilorLuxottica is actively pursuing commercialization of their Nuance Audio device in the US (Class 2 - OTC SaMD) and in the EU under the Class IIa classification for hearing aids. The device form factor is an eyeglass frame. Currently there are no medical devices marketed as a hearing aid in the intended form factor (Nuance Audio) which suggests the need for preclinical and clinical evaluations to assess any impact to non-clinical standards compliance and user clinical performance. The manufacturer is actively addressing standards compliance with qualified third-party laboratories and has engaged NAL to collaborate on the clinical assessments based on its extensive history and expertise in the personal hearing aid arena.

Clinical assessment of device performance (basic safety and effectiveness with intended users) will be conducted as per study protocol. Additionally, to ensure quality, preliminary bench top compliance testing will be conducted as part of the study prior to first participant enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Native English speakers
* Self-reported hearing or listening difficulties
* No need for prescription lenses (contact lenses acceptable)
* Ability to use smartphones and complete online surveys
* Willingness and ability to attend two in-person research appointments

Exclusion Criteria:

* Active ear disease, occluding cerumen, or any of the FDA "red flag" conditions
* Hearing asymmetry or sudden hearing changes
* Requirement for prescription eyewear (due to device form factor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2025-06-11 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
Speech intellegibility testing (Matrix test) with and without device | Day 1
  Conducted in both quiet and noise using validated Australian English BKB sentence materials.

SECONDARY OUTCOMES:
Real-world assessments | day 1
  Moderated walking tour in various acoustic settings (e.g., quiet rooms, traffic noise, multi-talker babble).

OTHER OUTCOMES:
Self-reported measures | Day 1
  Questionnaires assessing hearing difficulty (HHIE-S). The outcome measure is the grade of 10 questions ( 0 - 2 or 4 points per each question).
Self-reported measures | day 1
  Questionnaires assessing listening goals (COSI). The outcome measure is the grade in 5 different situation for entity of benefit ( on a scale from 1 to 5) and frequency of the benefit ( on a scale form 1 to 5)
Self-reported measures | day 1
  Questionnaires assessing perceived benefit (IOI-HA), The outcome measure is the grade to the questionnaire 7 questions on different scale ( raging from 1 to 5).

CONTACTS AND LOCATIONS:
Locations (1):
- National Acoustic Laboratories, Macquarie Park, New South Wales, Australia